CLINICAL TRIAL: NCT04230434
Title: Safety-Planning Intervention for Suicidal Behavior in an Emergency Department: an Effectiveness-implementation Hybrid Design
Brief Title: Implementability and Effectiveness of the Safety Planning Intervention for Suicidal Behavior
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto de Investigación Hospital Universitario La Paz (Other)
Collaborators: Hospital Universitario La Paz (Other); Fundacion para la Investigacion Biomedica del Hospital Universitario la Paz (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: SPI-EI
Record Dates: First submitted 2019-11-29; First posted 2020-01-18 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Suicide; Suicide, Attempted; Suicidal Ideation
Keywords: Suicide; Suicidal behavior; Suicidal attempt; Suicide prevention; Safety Planning Intervention
MeSH Terms: conditions — Suicide; Suicide, Attempted; Suicidal Ideation; Suicide Prevention

STUDY DESIGN:
Intervention Model Description: Interventional cohort (Safety Plan Intervention)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Safety Plan Intervention (Experimental): The Safety Plan Intervention (SPI) performed in ED or in ambulatory appointment
  Interventions: Behavioral: Safety Plan Intervention

INTERVENTIONS:
Behavioral: Safety Plan Intervention — The SPI has 6 key steps: (1) identify personalized warning signs for an impending suicide crisis; (2) determine internal coping strategies that distract from suicidal thoughts and urges; (3) identify family and friends who are able to distract from suicidal thoughts and urges and social places that provide the opportunity for interaction; (4) identify individuals who can help provide support during a suicidal crisis; (5) list mental health professionals and urgent care services to contact during a suicidal crisis; and (6) lethal means counseling for making the environment safer (Stanley & Brown, 2012)
  Other Names: Security Plan

SUMMARY:
The Safety Plan Intervention (SPI) has demonstrated to reduce suicide reattempts and to increase the ambulatory follow-up in american war veterans. This study evaluates the implementability and effectiveness in a significantly different population in a real world setting.

DETAILED DESCRIPTION:
We will perform a Effectiveness-implementation Hybrid Design (Curran et al. 2012) to study firstly the feasibility of implementing the SPI in our clinical setting and secondly its effectiveness. The experimental arm will consist in a group of patients who visit the ED for a suicide-related concern in which the SPI is performed. This will be in the Emergency Department , unless for clinical reasons, the ED psychiatrist decide to postpone it to the first psychiatric appointment (which will be before one week of the ED visit as part of the treatment as usual).

Right after the SPI is performed, both the patient and the clinician will complete questionnaire with satisfaction and acceptability measures. Subjects will be followed for 6 months. At this time medical records will be consulted to obtain suicide reattempts rates and follow-up adherence.

At all times, the anonymity of the participants will be preserved and will require heading of informed consent, as well as other ethical aspects indicated by the Ethics Committee.

ELIGIBILITY:
Inclusion criteria:

1. Suicide attempt or presence of severe suicidal ideation
2. Signed Informed Consent Form

Exclusion criteria:

1. Less than 18 years old
2. Hospitalization in the Psychiatry Department
3. Inability to understand the Safety Planning Intervention

Withdrawal criteria:

1) Participant's decision to withdraw from the trial

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2020-02-01 (Actual)

PRIMARY OUTCOMES:
Feasibility of Safety Plan Implementation | Baseline
  Percentage of SPIs performed in ED from total number of suicide related ED visits.

SECONDARY OUTCOMES:
Time required for the performance of the SPI | Baseline
  Minutes required for the performance of the SPI
Satisfaction of the patient with the Safety Plan | t0 (Safety Plan Performance )
  Likert-type scales with 5 levels of response will be measured through questions: "To what extent do the Safety Plan can help you to avoid a new situation of suicidal risk?"
Satisfaction of the Professional with the Safety Plan | Baseline
  Likert-type with 5 levels of response will be measured through questions: "To what extent do the Safety Plan can help you to avoid a new situation of suicidal risk?" Likert-type with 5 levels of response will be measured through questions: "To what extent the Safety Plan did you useful for the patient?". Open questions can be explained where contributions and obstacles encountered in its implementation will also be formulated.
Presence of suicide reattempt | Month 6
  Percentage of patients that commit suicide reattempt.
Time to suicide reattempt | Month 6
  Days from suicide attempt attended in the ED to the next suicide reattempt.
Adherence to psychiatric ambulatory follow-up | Month 6
  Percentage of patients that attend psychiatric ambulatory follow-up after ED discharge

OTHER OUTCOMES:
Predictive ability of the clinician in the subsequent conduct suicidal patient | Baseline
  is measured through a dichotomous question in which the professional will make a prognosis about the possibility that the patient may return to commit a suicidal behaviour.

CONTACTS AND LOCATIONS:
Overall Officials: Beatriz Rodriguez Vega, PhD, Principal Investigator — Instituto de Investigación Hospital Universitario La Paz
Locations (1):
- La Paz University Hospital, Madrid, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared with other researchers on request
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data will be available one year after publishing the final results for at least 5 years
Access Criteria: Please contact PI Beatriz Rodríguez-Vega (beatrizrvega@gmail.com)